CLINICAL TRIAL: NCT00845702
Title: Evaluation of Dotarem-enhanced Magnetic Resonance Angiography (MRA) Compared to Time-Of-Flight (TOF) MRA in the Diagnosis of Renal Arterial Disease
Brief Title: Renal Magnetic Resonance Angiography (MRA) Study Comparing Dotarem and Time Of Flight (TOF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment.
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-046
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Renal Artery Stenosis
Keywords: Renal artery stenosis; Contrast agent; MRA
MeSH Terms: conditions — Renal Artery Obstruction | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dotarem (Experimental): Each subject will receive one injection of Dotarem 0.2 ml/kg.
  Interventions: Drug: Gadoterate meglumine (Dotarem)
- Time Of Flight Magnetic Resonance Angiography (Other): Each subject undergo a TOF MRA
  Interventions: Other: Time of Flight Magnetic Resonance Angiography

INTERVENTIONS:
Drug: Gadoterate meglumine (Dotarem) — Each subject will receive one injection of Dotarem 0.2 ml/kg
  Arms: Dotarem
Other: Time of Flight Magnetic Resonance Angiography — Each subject will undergo a TOF MRA
  Arms: Time Of Flight Magnetic Resonance Angiography

SUMMARY:
The study will evaluate the efficacy and safety of Dotarem enhanced MRA compared to TOF MRA in patients suffering from renal arterial disease.

DETAILED DESCRIPTION:
Each participant will undergo first a TOF MRA followed by a Dotarem-enhanced MRA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged more than 18 years,
* Strongly suspected of having renal arterial disease,
* Scheduled (or to be scheduled) to undergo arterial catheter-based X-ray angiography examination,

Exclusion Criteria:

* Known grade IV or V chronic kidney disease (GFR<30 mL/min/1.73m²),
* Contraindication to MRI,
* Acute renal dysfunction within the 6 months preceding Dotarem®-enhanced MRA examination,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Guerbet LLC, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit: Apr 2009 Last Patient Last Visit: Feb 2010 Location: Radiology centers
Pre-assignment Details: Out of the 33 enrolled patients, one patient did not undergo any of the planned procedures due to an inability to obtain an intravenous access with the initial planned procedure.
Groups:
- TOF Followed by Dotarem-enhanced MRA: Each patient will undergo a Time-Of-Flight Magnetic Resonance Angiography followed by an Dotarem-enhanced Magnetic Resonance Angiography(with an injection of Dotarem 0.2 ml/kg).
Period: TOF MRA
Arm/Group | TOF Followed by Dotarem-enhanced MRA
Started | 33
Completed | 32 (One patient did not perform study MRA procedures.)
Not Completed | 1
Period: Dotarem MRA
Arm/Group | TOF Followed by Dotarem-enhanced MRA
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures were recorded for all 33 patients.
Groups:
- TOF and Dotarem Enhanced MRA: Each subject will undergo a Time of Flight Magnetic Resonance Angiography followed by a Dotarem-enhanced Magnetic Resonance Angiography (with injection of Dotarem 0.2 ml/kg).
Arm/Group | TOF and Dotarem Enhanced MRA
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Percent of Non Assessable Renal Artery Segments
Description: For each examination (TOF and Dotarem MRA) the percent of non-assessable segment will be compared
Time Frame: 1 to 7 days
Population: The study has been prematurely terminated, and the planned analyses were not done
Groups:
- Dotarem MRA: Each subject will receive one injection of Dotarem 0.2 ml/kg.
- Time Of Flight MRA: Each subject will undergo a TOF MRA
Arm/Group | Dotarem MRA | Time Of Flight MRA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Dotarem Magnetic Resonance Angiography: Each subject will receive one injection of Dotarem 0.2 ml/kg.
- Time Of Flight MRA: Subjects undergo a TOF MRA
Arm/Group | Dotarem Magnetic Resonance Angiography | Time Of Flight MRA
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/32
Other Adverse Events (participants affected / at risk) | 6/32 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem Magnetic Resonance Angiography (N=32) | Time Of Flight MRA (N=32)
Mental status changed (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem Magnetic Resonance Angiography (N=32) | Time Of Flight MRA (N=32)
Investigation (Investigations) | 3 (3) | 0 (0)
General disorders (General disorders) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was not completed due to poor enrollment. The statistical analysis was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days